



EHSREC No: 2024\_06\_02

#### **DETAILED VOLUNTEER INFORMATION SHEET**

#### Dear Volunteer,

We are carrying out a study on the experiences of hospital-based doctors and nurses across the EU. This information sheet will tell you what the study is about.

### What is the study about?

As part of an EU funded KEEPCARING project (101137244) the study aims to find out what are the current risks and levels of burnout among hospital-based doctors and nurses in the EU and how do factors like work setting, leadership and resilience influence it, and what the health services can do about it.

### **KEEPCARING Project**

This survey is part of a larger research project, KEEPCARING, funded by the EU (grant no. 101137244). The KEEPCARING project aims to address the stress and burnout among healthcare professionals in the European Union. Healthcare professionals, especially those working in hospital settings, face extraordinary levels of stress and pressure. The COVID-19 pandemic further intensified these stressors, revealing systemic vulnerabilities in healthcare systems across Europe. While some interventions to improve wellbeing and resilience exist, there is still a significant gap in understanding what combination of solutions works best, especially in high-stress, surgical environments.

The KEEPCARING project was initiated with the goal of fundamentally improving the well-being of healthcare professionals across the European Union. The project seeks to co-create a comprehensive solution package specifically designed to reduce stress and enhance resilience in healthcare workers at every level—individuals, teams, and organizations. This study is the first stage of the project, which includes finding the levels of burnout, what factors hinder and support it, such as work environment, leadership, and resilience. Further details about KEEPCARING can be found here.

### What are the benefits of participating in the survey?

We hope that you will benefit as a participant by having a space to share your knowledge and experience and have your voice heard.

However, in particular, the findings of the study will help raise awareness of the levels of burnout among hospital-based doctors and nurses working at the coalface. A snapshot of the findings will be made available to your relevant associations/organisations so they can also raise awareness of these burnout levels.

Other potential benefits include.

- Contributing to development of best management and intervention practices to manage burnout in hospital nursing and medical staff.
- New empirical research that will drive innovation on addressing burnout in hospital-based doctors and nurses.

#### What are the risks?

You might decide that you do not want to answer a question. If this happens, you do not have to answer any question you do not wish to. If you get upset and need support, we will be happy to signpost you to support services.

As with all research surveys/interactions, there are data protection and privacy risks. The survey is administered through a University of Limerick approved Qualtrics account. Please note, your IP address may be collected once you complete the survey, but this will be deleted when we transfer the data from Qualtrics for analysis. The University has invested in commercial Microsoft accounts which have the highest level of security, and if you ticked the box for the interview part this will also be done on MS Teams and is also secure. All the Universities' policies and procedures for IT security and data protection will be followed.

### What if I do not want to take part?

Participation in this study is completely voluntary and you can choose whether or not to take part. You can stop your involvement in the survey at any time simply by exiting the survey.

## What happens to the information?

Please note, that while we do not collect direct identifiers about you, if you provide your email address we will be able to link your answers with your email address. Be assured however, that all the information that is collected will be kept private including your email address and stored securely and safely on the researchers' University of Limerick's One Drive. All our devices are encrypted, and also protected with a password, anti-virus software and VPN.

For future studies using non-invasive biomarkers such as heart rate variability and breathing rate, we aim to link your survey responses to this data, and your email address will be deleted after research partner responsible for this part of the project, Universidade NOVA de Lisbia, contacts you. In case of the interview study, your email address will be deleted after we contact you in relation to that study.

All email addresses will be deleted after 36 months. The data that is gathered in the study will be kept for seven years. After this time, it will be destroyed. We have also included a link to our Research Privacy Notice which has more information as to what happens to your information.

### Who else is taking part?

Doctors and nurses, as well as trainee doctors and nurses aged 18 or over from several EU countries including Ireland, Germany, Denmark and the Netherlands.

### What if something goes wrong?

It is unlikely that something will go wrong during the survey. Possible scenarios: poor connection or loss of internet connection.

## What happens at the end of the study?

At the end of the study the information will be used to present results, including in academic forums such as journal articles and conferences. The researcher has agreed a plan to communicate the results to any of the support organisations that sent out the study information including providing a copy to any pre-print article. A copy of the written research paper will be freely available through the UL repository, and the link to this will be published on social media including your support organisations.

Anonymised data from data collection will be made available to used by in academic papers, conference presentations and posters, and other academic forums. This may also be used in other communications to share the results such as blog posts, newsletter articles. No names or any participant identifiers, or third parties names will appear in any of the results or communication materials.

As mentioned above, this study is part of a wider EU-funded project KEEPCARING (see partners below) on burnout in healthcare workers in EU countries, therefore, after being anonymised, the data collected will be shared with the other data controllers - partners of the project (Universidade NOVA de Lisboa, Portugal, University of Coimbra, Portugal, Copenhagen University Hospital, Rigshospitalet, Denmark, and Universitätsklinikum Hamburg-Eppendorf, Germany.

We are also subject to the policies and procedures of University of Limerick (UL) and the EU Commission. As an institution, UL and EU commission are committed to Open Science. This means that anonymised data sets (such as anonymous survey data sets) may be made available to other researchers following a strict set of guidance criteria.

# What if I have more questions or do not understand something?

If you have any questions about the study, you may contact stephen.gallagher@ul.ie. It is important that you feel that all your questions have been answered at any stage during the research process.

### How do I take part?

You can take part by following the link to the survey here or using the QR code to access it.

#### **Contact information of Project Investigators:**

# **Principal Investigator**

Prof. Stephen Gallagher, Dept of Psychology. University of Limerick, Tel (061) 234899 Email: Stephen.Gallagher@ul.ie

#### **Co-Investigators**

Dr. Trina Tamrakar and Melissa Blunnie, Department of Psychology. University of Limerick,

Email: Trina.Tamrakar@ul.ie

Thank you for taking the time to read this. We would be grateful if you would consider participating in this study.

Please click here to go back to the survey.

This research study has received Ethics approval from the Education and Health Sciences Research Ethics Committee [2024\_06\_02].

If you have any concerns about this study and wish to contact someone independent, you may contact:

Chair Education and Health Sciences Research Ethics Committee EHS Faculty Office University of Limerick Tel (061) 234101

Please click here to go back to the survey.